CLINICAL TRIAL: NCT02399865
Title: A Randomised Controlled Trial of Family and Social Network Intervention for Young People Who Misuse Alcohol and Drugs: a Feasibility Study [Y-SBNT]
Brief Title: Family and Social Intervention for Young People
Acronym: YSBNT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: University of York (Other); Birmingham and Solihull Mental Health NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Northumberland, Tyne and Wear NHS Foundation Trust (Other); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIHR 11/60/01
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Alcohol Misuse; Drug Misuse
MeSH Terms: conditions — Drug Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- YSBNT Group (Experimental): Six 50 minute YSBNT sessions (delivered by a trained YSBNT practitioner) for over a maximum period of 12 weeks
  Interventions: Other: Youth Social Behaviour and Network Therapy
- Treatment as Usual Group (No Intervention): Usual care delivered by treatment-as-usual practitioners

INTERVENTIONS:
Other: Youth Social Behaviour and Network Therapy — The Y-SBNT will be delivered according to the developed purpose-designed therapy manual. Participants randomised to Y-SBNT will be offered six, 50 minute SBNT sessions for over a maximum period of 12 weeks. Where consent is obtained, sessions will audio-recorded and reviewed by the research team to ensure fidelity with the YSBNT manual and principles of practice.
  Using the identification of the social network of the young person conducted in the first session as a platform, subsequent core strategies of the adapted YSBNT approach include motivational techniques, improving communication and coping mechanisms, and crucially given the nature of substance misuse, developing a network-based relapse management plan. Participants will be given the opportunity to invite members of their network to the treatment sessions. The therapeutic approach also has scope to address client-focussed elective areas, for example, educational requirements.
  Other Names: YSBNT
  Arms: YSBNT Group

SUMMARY:
Research evidence shows that there is a high prevalence of substance use among young people in the UK. Early onset and high levels of use are associated with a range of negative outcomes, including increased risk of later problematic use and dependence. A growing body of research has identified family interventions to be effective in treating young people's substance use problems. However, despite this evidence, takeup of family based approaches, at least in the UK, has been low. A key factor appears to be the resource intensive nature of many family interventions, making them difficult to implement and deliver in many service settings, especially in the context of substantial cuts to drug and alcohol services for young people (1). Another potential barrier may be the cultural adaptation of approaches developed in the USA to a UK setting. There is growing awareness of the need to adapt evidence-based treatments to different cultural groups and settings in order to ensure successful implementation (2,3,4).

Following on from developmental and adaptation work, this study aims to demonstrate the feasibility of recruiting young people to specifically developed family and network based intervention. In addition the feasibility of training staff from existing young people addiction services to deliver this intervention will be explored and treatment retention will be assessed. Qualitative interviews will elicit the participants' views on the acceptability of the intervention and their experiences of both it and the study process.

DETAILED DESCRIPTION:
Following the adaptation, we developed a manualised family-based intervention for young substance misusers up to the age of 18. This was an evidence-based approach, drawing on our previous research, a review of the literature and the views of young substance misusers with experience of treatment (Phase 1).

We aim to undertake a smallscale trial in two sites (Phase 2), to assess both the feasibility of the intervention and the scope for moving to a full trial of clinical and cost effectiveness. We also aim to evaluate the implementation of this new intervention using mixed methods research , monitoring randomisation procedures, treatment fidelity, staff time (and associated costs), engagement, retention and a range of outcome measures, reflecting the multiple vulnerabilities of this population. We will thereby address the brief's central aims of assessing the feasibility of a familybased intervention with this group and whether a trial could be successfully undertaken.

Phase 1: Intervention Development Using the original Intervention structure and content as a platform, the overall aim was to adapt this family and social intervention in collaboration with those who have experience of using services in order to ensure that it is acceptable to young people and their families, remains focused on the important aspects that promote and support behaviour change and yet is realistic and deliverable in a way that maximises treatment engagement, taking into account young people's views and preferences. The resulting intervention will therefore be one in which much of the original material is oriented to a youth population, whilst retaining the key principles of the original Social Behaviour and Network Therapy. At the time of completing this ethics application, two of the three key sources of information which informed this process were already carried out. First, a Systematic Review was conducted on the already existing evidencebase on the effectiveness and acceptability of family based interventions in treating young people's substance abuse. Second, Patient and Public Involvement (PPI) was carried out by actively engaging a sample of young people with a history of treatment for substance abuse in a number of consultation processes. Third, we are yet to explore the the point of view of those who will deliver the intervention by drawing on a group of therapists and service managers working in child and adolescent addiction services. This group will comment on each stage of the intervention and handbook design, being invited to 'walk through' the delivery of this new intervention.

Phase 2: Feasibility Randomised Controlled Trial (RCT) The purpose of this ethics application is to obtain ethical approval for this specific phase of our study. For phase 2 we propose a prospective pragmatic randomised controlled trial to assess the feasibility and impact of the adapted family and social network intervention for drug and alcohol misuse in young people. The proposed trial will use concealed randomisation, intention to treat analysis and characterisation of refusers and dropouts. It will be a pragmatic trial, delivered in two Young People services. It involves a parallel group design comparing two conditions: (i) Adapted youth social network intervention (YouthSBNT) and (ii) Treatment as usual.

For those that agree to participate, the researcher will:

1. Obtain written consent from them to participate in the trial;
2. Conduct a baseline assessment;
3. Telephone the York Trials Unit Freephone randomisation service or use the online system to randomise the patient (hereafter referred to as the participant);
4. Provide the participant with an appointment to see the therapist or clinician appropriate to their allocation.

At baseline, information will be collected from the patient regarding their drug and alcohol use, emotional wellbeing, social network, family environment, quality of life, school attendance, selfreported crime, health care use, social services contact, and demographics. The same set of information will be collected at 3 months and 12 months follow up postrandomisation assessments. Interviews will be undertaken by the research fellows, covering the main and secondary outcome measures mentioned earlier. In addition, qualitative interviews will be used to explore the acceptability and wider context of the impact of the intervention to the young people and their family members/social network. Economic evaluation will also be conducted to inform larger definitive trial.

ELIGIBILITY:
Inclusion Criteria:

(i) Young people with drug and/or alcohol problems newly referred and accepted for treatment by the two agencies during the period of recruitment. (ii) Willing to provide written informed consent. (iii) Able to provide written informed consent.

Exclusion Criteria:

(i) Concurrent severe mental illness that precludes them from active participation.

(ii) Severe physical illness that precludes them from active participation. (iii) Unable or unwilling to give written informed consent.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 3 months
  Quantitative assessment of the acceptability of the research will be assessed by numbers referred, number eligible and those agreeing to participate.
Retention in Treatment | 3 months (12 weeks)
  Retention in treatment will be evaluated by number of sessions attended as a measure of acceptability of the interventions to participants.
Follow up completion rates | 12 months
  Quantitative assessment of the number of follow-up interviews completed.

SECONDARY OUTCOMES:
Qualitative Interviews | 3 to 12 months
  The acceptability of the Y-SBNT intervention to the young people and the wider context of the impact of the intervention will be explored by undertaking semi-structured qualitative interviews conducted at three and 12 months post-randomisation. In addition, the acceptability of the intervention to those attending as network members will be explored through similarly semi-structured interviews at three months post-randomisation.
Emotional Well-being as measured by Social Difficulties Questionnaire (SDQ) | 12 months
  Emotional well-being will be measured at baseline, three and 12 months post-randomisation using the Strengths and Difficulties Questionnaire (SDQ) has five separate sub-scales for different aspects of problems or behaviours: emotional problems, conduct/behaviour problems, inattention/hyperactivity, relationships with peers, and pro-social behaviour. The first four scales can be added together to produce a score for total difficulties. The SDQ has been used extensively and has demonstrated high levels of reliability and validity
Social Network Support as measured by Important People Drug and Alcohol interview (IPDA) | 12 months
  Given the emphasis on family and peer support of the intervention, social network support will be measured at baseline, three and 12 months post-randomisation using the IPDA in order to understand the influence of social support on treatment for substance misuse. Researchers have described 4 sub-types of support: General structural support refers to embeddedness in a social network. e.g. number of close friends; Abstinence-specific structural support is the prevalence of nondrug or alcohol users relative to drug or alcohol users in the social network; General functional support refers to assistance from others that does not specifically address drug or alcohol use (e.g. giving advice); Abstinence-specific functional support consists of behaviours that focus on abstinence or substance use more directly, such as encouraging someone to remain in treatment or (as a negative example) offering alcohol or drugs. These four areas will be covered using the IPDA.
Family Environment as measured by Family Environment Scale (FES) | 12 months
  Family environment will be measured at baseline, three and 12 months post-randomisation using the 27-item Relationship dimension of the FES consisting of Cohesion, Expressiveness, and Conflict subscales (9 items each). It is designed to measure the atmosphere in the family household and will be used where appropriate to the circumstances of the participant. These subscales measure support, expression of opinions, and angry conflict within a family. This 27-item measure has been used by some of the applicants in previous studies and yields scores for family cohesion, free expression of emotion in the family and absence of open conflict.
Working Alliance Inventory | 3 months
  Working Alliance Inventory will be administered at end of treatment sessions one and three to the young people and also to the therapists delivering the intervention and treatment as usual. The questionnaire measures the perceived strength of the working alliance between therapists and their clients during therapy sessions. The young people will be provided with envelopes to seal their completed WAI in.
Health Related Quality of Life (HRQoL) | 12 months
  HRQoL will be assessed at baseline, three and 12 months post-randomisation using the European Quality of Life - 5 Dimensions-5 levels (EQ-5D-5L). EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal, where health is characterised on five dimensions (mobility, self-care, ability to undertake usual activities, pain, anxiety / depression).

OTHER OUTCOMES:
Activities and Engagement | 12 months
  School attendance and engagement; self-reported crime and health care and social services contact will be measured at baseline and 12 months post-randomisation.
Intervention effectiveness as measured by Timeline Follow-Back (TLFB) | 90 days
  This outcome measure will be based on the TLFB interview and will be the proportion of days on which the main problem substance was used in the preceding 90 day period covered by each assessment point (baseline, 3 and twelve months post-randomisation).
Young peoples' involvement | 24 months
  This study will allow us to explore ways in which young people with experience of using services can be involved in a study of this nature, informing patient and public involvement (PPI) in a larger trial that may take place. Learning from the study will also contribute to the wider emerging evidence base on PPI, and hopefully inform other studies and involvement activity with young people whose voices are less frequently heard, or who may be excluded by traditional models of patient and public involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Alex G Copello, PhD, Principal Investigator — University of Birmingham

REFERENCES:
- [Background] 1.Drugscope. Charities warn of 'devastating impact' of cuts to young people's drug and alcohol services. 2011; 20 July. 2.Bernal G, JimenezChafey M, Domenech Rodriquez MM. Cultural adaptation of treatments: a resource for considering culture in evidencebased practice. Professional Psychology; Research and Practice. 2009: 40 (4); 361368. 3.Cortese CA (1999). Drug services and cultural adaptation. Drugs: education, prevention and policy. 1999: 6 (3); 361366 4.Lau, A.S. Making the case for selective and directed cultural adaptations of evidence-based treatments: examples from parent training. Clin Psychol Sci Prac. 2006: 13; 295310.
- See also: Protocol paper published in Pilot and Feasibility Studies — http://www.pilotfeasibilitystudies.com/content/1/1/8